CLINICAL TRIAL: NCT04464031
Title: Study on the Application Value of Electronic Alert for Acute Kidney Injury in Geriatric Wards
Brief Title: Electronic Alert for Acute Kidney Injury in Geriatric Wards
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20181015
Record Dates: First submitted 2020-06-16; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-06

CONDITIONS: Acute Kidney Injury
Keywords: Acute kidney injury; Alert; Geriatric wards
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alert group (Experimental)
  Interventions: Other: electronic alert
- Control group (No Intervention)

INTERVENTIONS:
Other: electronic alert — The e-alert system was developed by the divisions of Nephrology and Information Management of Guangdong Provincial People's Hospital (Patent Application 201610001950.5). The alert system made a diagnosis of acute kidney injury according to Kidney Disease: Improving Global Outcomes criteria. Then, the doctor receives an alert of acute kidney injury.
  Arms: Alert group

SUMMARY:
Operating acute kidney injury electronic alert in geriatric wards; Acute authenticity evaluation of acute kidney injury electronic alert; To explore the clinical value of electronic alert for acute kidney injury prevention and treatment in geriatric wards.

ELIGIBILITY:
Inclusion Criteria:

* Age over 65 years old
* Diagnose of acute kidney injury by e-alert

Exclusion Criteria:

* Baseline serum creatinine > 4mg/dL
* Stage-5 chronic kidney disease or maintenance hemodialysis
* Kidney transplantation
* Amputation

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis rate of acute kidney injury (Rate of missed diagnosis); | 1 year
Rate of dialysis | 1 year
Rate of death | 1 year

SECONDARY OUTCOMES:
Rate of nephrology consultation | 1 year
Rate of nephrology follow-up | 1 year
Renal function after 90 days of acute kidney injury | 1 year

IPD SHARING:
Plan to Share IPD: No